CLINICAL TRIAL: NCT00632398
Title: Couples and Cancer: Building Partner Efficacy in Caring
Brief Title: Multimedia Training for Family Caregivers in Use of Touch and Massage in Supportive Cancer Care
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Collinge and Associates, Inc. (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, William Collinge, PhD, President, Collinge and Associates, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000587451; COLLINGE-06-200
Record Dates: First submitted 2008-03-07; First posted 2008-03-10 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Cancer
Keywords: massage; oncology massage; palliative care; supportive care; integrative oncology; informal caregiving; spouse caregiving; family caregiving; caregiver education; psychosocial oncology; caregiver stress; coping with cancer; quality of life; end of life care
MeSH Terms: conditions — Neoplasms; Caregiver Burden | interventions — Touch

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention control (reading) (Active Comparator): Caregivers read to patients from literature of the patient's choice for recommended 20 minutes at least 3 times per week for 4 weeks.
  Interventions: Behavioral: Attention control (reading)
- Touch, Caring and Cancer DVD program (Experimental): Caregivers apply the instruction of the Touch, Caring and Cancer DVD program for patients for recommended 20 minutes at least 3 times per week for 4 weeks.
  Interventions: Behavioral: Touch, Caring and Cancer DVD program

INTERVENTIONS:
Behavioral: Attention control (reading) — Caregivers read to the patient from literature of the patient's choice for recommended 20 minutes at least 3 times per week for 4 weeks
  Arms: Attention control (reading)
Behavioral: Touch, Caring and Cancer DVD program — DVD- and manual-based instruction for caregivers and patients in the use of touch and massage techniques as supportive care in cancer, including: preparation for a session, safety precautions related to cancer and its treatments, communication about touch, centering to calm the mind; manual techniques for the head, neck, shoulders, back, feet and hands to promote relaxation; and acupressure for pain, nausea and anxiety.
  Arms: Touch, Caring and Cancer DVD program

SUMMARY:
RATIONALE: A multimedia education program for family caregivers that teaches simple methods of touch and massage for the comfort of cancer patients at home may be effective in lowering stress, reducing symptoms, and improving quality of life for patients; and may improve caregiver satisfaction and self-efficacy.

PURPOSE: This randomized phase II trial is studying how well multimedia instruction of caregivers in use of touch and massage works for cancer patients and their care partners.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Produce a multimedia program to deliver instructional content in massage for cancer patients and their lay care partners.
* Determine the effects of the multimedia program on care partner esteem and stress and on the frequency and duration of the care partner's provision of their assigned form of support to the patient.
* Determine the effects of the multimedia program on patient symptom levels, functional quality of life, perceived stress, and physiologic indices of stress.

Secondary

* Examine the impact of the multimedia program on care partner concerns about use of touch as a form of support, and on self-efficacy in massage.

OUTLINE:

* Multimedia program production and screening (year 1): Patient/care partner dyads representative of a broad spectrum of relationships participate in filming a multimedia program about massage, acupressure, light touch, and massage safety precautions. The multimedia program is titled, "Massage for People with Cancer: Simple Instruction for Family and Friends." The program comprises a menu-driven DVD which allows the viewer to select English or Spanish as well as individual chapters of content, and a manual keyed to the DVD content. A different set of diverse patient/care partner dyads screen and critique the multimedia program.
* Randomized controlled study of program's efficacy (year 2): Patient/care partner dyads who reside in the same home are recruited. Dyads within each race/ethnic group are stratified by patient total scores on the baseline FACT-G assessment. Dyads are then randomized to 1 of 2 arms.

  * Arm I (experimental intervention): Dyads attend an orientation meeting with other dyads of their language group in order to meet the Oncology Massage Therapist (OMT) and research assistant (RA) assigned to them during the study; watch the DVD together and discuss it afterward; receive instructions for weekly data collection; and receive explanation about the safety monitoring home visit and the bi-weekly phone monitoring. Instructions for data collection include instructions for the care partner to fill out a sample of the weekly Study Report card. Dyads are given the DVD and manual to take home, and those who do not have a DVD player are provided one. Dyads complete at least one massage over at least 20 minutes once a week for 20 weeks in which they provide the techniques demonstrated in the film. An OMT makes a home visit to each dyad during the first 2 weeks, and then as needed, to monitor for understanding of and adherence to the relevant safety precautions for the given patient. Dyads receive bi-weekly telephone monitoring from an RA in order to encourage compliance with the weekly activity and monitor for any adverse events or safety concerns that warrant another home visit by the dyad's OMT (e.g., changes in medical treatment that call for changes in precautions).
  * Arm II (control intervention): For 4 weeks, care partners spend at least 20 minutes a week alone with the patient, reading to the patient from literature of interest to the patient. The literature may be fiction, non-fiction, or poetry that does not contain news or stressful subject matter. Dyads receive telephone monitoring from their RA within the first week and then every 2 weeks thereafter to encourage compliance, monitor for any adverse events or concerns, and respond to questions about the project. At the end of the 4 weeks, dyads attend an orientation meeting with the Principal Investigator, OMTs, and RAs. At this meeting, dyads view the multimedia program and discuss precautions and any other issues that may affect their utilization of the instruction. Dyads are then given the multimedia program to take home, and a DVD player if they need one. A home visit by an OMT is scheduled to assure the dyad understands and implements relevant safety precautions. The dyads then participate in the use of the intervention for the remaining 16 weeks of the study.

All participants in the study complete quality of life, perceived stress, and other questionnaires at baseline and then at 4, 12, and 20 weeks. Demographic and patient medical information is also collected. Saliva samples are collected from patients at baseline and then at 4, 12, and 20 weeks to monitor cortisol and DHEA levels.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cancer patient and their care partner with any of the following characteristics:

  * African American
  * Asian
  * Hispanic or Latino
  * Caucasian
  * Intimate relationship
  * Parent/adult child relationship
  * Same-sex couple relationship
  * Male or female
* Patient must have undergone conventional cancer treatment within the past 6 months

PATIENT CHARACTERISTICS:

* Speaks, reads, and writes English, Spanish, or Chinese (care partner)
* Speaks, reads, and writes English, Spanish, or Chinese (patient)
* No contraindication, such as serious mental illness or physical inability, that would preclude study participation (patient or care partner)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Acute effects of massage on patient symptoms as assessed by the weekly Study Report card
Longitudinal effects of massage on patient symptoms as assessed by the weekly Study Report card
Frequency and duration of care partner providing the assigned form of support as assessed by the weekly Study Report card
Care partner esteem as assessed by a 7-item esteem subscale of the Caregiver Reaction Assessment at baseline and then at 12 and 24 weeks
Patient physiological stress measures as assessed by measuring diurnal variation in cortisol and DHEA at baseline and then at 12 and 24 weeks
Patient and care partner perceived stress as assessed by the Perceived Stress Scale at baseline and then at 12 and 24 weeks
Patient functional quality of life as assessed by FACT-G at baseline and then at 12 and 24 weeks

SECONDARY OUTCOMES:
Care partner self-efficacy and concerns about using touch as support as assessed by an investigator-generated survey at baseline and then at 12 and 24 weeks
Care partner utilization of multimedia materials as assessed by the weekly Study Report card

CONTACTS AND LOCATIONS:
Overall Officials: William Collinge, PhD, MPH, Principal Investigator — Collinge and Associates, Inc.
Locations (3):
- United States (3):
  - Collinge and Associates, Kittery, Maine
  - Greater Boston Chinese Golden Age Center, Boston, Massachusetts
  - Latin American Health Institute, Boston, Massachusetts

REFERENCES:
- [Background] Collinge W, MacDonald G, Walton T. Massage in supportive cancer care. Semin Oncol Nurs. 2012 Feb;28(1):45-54. doi: 10.1016/j.soncn.2011.11.005. PMID 22281309
- [Result] Collinge W, Kahn J, Walton T, Kozak L, Bauer-Wu S, Fletcher K, Yarnold P, Soltysik R. Touch, Caring, and Cancer: randomized controlled trial of a multimedia caregiver education program. Support Care Cancer. 2013 May;21(5):1405-14. doi: 10.1007/s00520-012-1682-6. Epub 2012 Dec 21. PMID 23262808